CLINICAL TRIAL: NCT00978679
Title: Peripheral Refraction and Aberration in Myopic Progression and Myopic Control
Brief Title: Peripheral Optics in Myopia and Orthokeratology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Menicon Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Pauline Cho, Professor, The Hong Kong Polytechnic University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-RGVM
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Myopia
Keywords: Children; Peripheral refraction; Aberration; Eyeball length; Myopic control; Myopia; Corneal reshaping; Orthokeratology
MeSH Terms: conditions — Myopia | interventions — Eyeglasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orthokeratology (Experimental): Myopic children wearing orthokeratology at night will be the study group
  Interventions: Device: Orthokeratology lenses
- Others (Other): Myopic children wearing single-vision spectacles in the daytime will serve as control group
  Interventions: Device: Spectacles

INTERVENTIONS:
Device: Orthokeratology lenses — Nightly use of orthokeratology lenses to correct the refractive errors
  Other Names: Menicon Z Night Lens 2; Menicon Z Night Lens 2 Toric
  Arms: Orthokeratology
Device: Spectacles — Daily use of single vision lenses to correct refractive errors
  Other Names: Glasses; Eyeglasses
  Arms: Others

SUMMARY:
The primary objective of the current study is to investigate changes in peripheral refraction and aberration in children wearing orthokeratology lenses and single-vision spectacles.

DETAILED DESCRIPTION:
Apart from being effective in reducing low to moderate myopia, orthokeratology has been shown to have potential in retarding myopic progression. The central cornea is flattened and peripheral optics altered in orthokeratology and it has been suggested that orthokeratology slows myopic progression through the alteration of peripheral optics. The aim of the current study is to investigate the changes in peripheral refraction and aberration in children wearing orthokeratology (study group) and single-vision spectacles (control group).

ELIGIBILITY:
Inclusion Criteria:

* Myopia (refractive sphere): > 0.50D and ≤ 6.00D
* Astigmatism: with-the-rule astigmatism (axes 180 +/- 30) ≤ 1.50D; astigmatism of other axes ≤ 0.50D
* Spherical equivalent (SE): > 0.50D and ≤ 6.75D (myopia)
* Best corrected monocular visual acuity: equal to or better than 6/7.5 in Snellen scale
* Willingness to wear contact lenses or spectacles on a daily basis
* Availability for follow-up for at least 2 years

Exclusion Criteria:

* Strabismus at distance or near
* Contraindication for contact lens wear and orthokeratology (e.g. limbus to limbus corneal cylinder and dislocated corneal apex)
* Prior experience with the use of rigid lenses (including orthokeratology)
* Prior experience with myopic control treatment (e.g. refractive therapy or progressive spectacles)
* Systemic or ocular conditions which may affect contact lens wear (e.g. allergy and medication)
* Systemic or ocular conditions which may affect refractive development (e.g. Down syndrome, ptosis)

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2008-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in cycloplegic off-axial auto-refraction, aberration and eyeball length | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Cho, PhD, Principal Investigator — School of Optometry, The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, The Hong Kong Polytechnic University, Hong Kong, Hong Kong, China

REFERENCES:
- [Background] Mathur A, Atchison DA. Effect of orthokeratology on peripheral aberrations of the eye. Optom Vis Sci. 2009 May;86(5):E476-84. doi: 10.1097/OPX.0b013e31819fa5aa. PMID 19342979
- [Result] Cho P, Cheung SW, Edwards M. The longitudinal orthokeratology research in children (LORIC) in Hong Kong: a pilot study on refractive changes and myopic control. Curr Eye Res. 2005 Jan;30(1):71-80. doi: 10.1080/02713680590907256. PMID 15875367
- [Result] Walline JJ, Jones LA, Sinnott LT. Corneal reshaping and myopia progression. Br J Ophthalmol. 2009 Sep;93(9):1181-5. doi: 10.1136/bjo.2008.151365. Epub 2009 May 4. PMID 19416935
- [Result] Charman WN, Mountford J, Atchison DA, Markwell EL. Peripheral refraction in orthokeratology patients. Optom Vis Sci. 2006 Sep;83(9):641-8. doi: 10.1097/01.opx.0000232840.66716.af. PMID 16971842